CLINICAL TRIAL: NCT06786390
Title: Regaining Walking Ability Easier and Better in Critical Illness Polyneuropathy and Myopathy
Brief Title: Improved Recovery of Walking in Acquired Muscle Weakness
Acronym: Re-Walk-Easy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Re-Walk-Easy-SC
Record Dates: First submitted 2024-12-19; First posted 2025-01-22 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Critical Illness Myopathy; Critical Illness Polyneuropathy
Keywords: Functional Electrical Stimulation; Acquired Muscle Weakness; Rehabilitation
MeSH Terms: conditions — Polyneuropathies | interventions — proto-oncogene protein c-fes-fps

STUDY DESIGN:
Intervention Model Description: A double-blind longitudinal RCT will be performed. The subjects enrolled will be divided in two groups on the basis of their diagnosis, CIP/CIM. Subsequently subjects will be randomly assigned either to the experimental group (FES), or to the control group (CON).
Who Masked: Participant, Outcomes Assessor
Masking Description: Researchers devoted to data collection and Patients will be masked to the allocated treatment. On subjects belonging to control group, the stimulation device will be placed normally and the stimulation intensity will be set at 0.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CIP-FES (Experimental): Each subject will receive 15 individual rehabilitation sessions, each lasting 60 minutes, conducted 3 to 5 times per week over a period of 5 to 3 weeks, depending on the weekly frequency,
  Intentional, repetitive movements, such as lower limb movements within goal-oriented mobility tasks, will be performed, with FES applied in parallel. Two approaches will be used: (i) assistive stimulation for passive patients with poor muscle strength, and (ii) proportional active stimulation for subjects with residual muscle strength.
  Interventions: Other: Rehabilitation protocol: FES
- CIM-FES (Experimental): Each subject will receive 15 individual rehabilitation sessions, each lasting 60 minutes, conducted 3 to 5 times per week over a period of 5 to 3 weeks, depending on the weekly frequency,
  Intentional, repetitive movements, such as lower limb movements within goal-oriented mobility tasks, will be performed, with FES applied in parallel. Two approaches will be used: (i) assistive stimulation for passive patients with poor muscle strength, and (ii) proportional active stimulation for subjects with residual muscle strength.
  Interventions: Other: Rehabilitation protocol: FES
- CIP-CON (Active Comparator): Each subject will receive 15 individual rehabilitation sessions, each lasting 60 minutes, conducted 3 to 5 times per week over a period of 5 to 3 weeks, depending on the weekly frequency,
  Intentional, repetitive movements, such as lower limb movements within goal-oriented mobility tasks (e.g., overground straight walking), will be performed without FES. The electrical stimulator will be positioned, and the amplitude will be set to zero
  Interventions: Other: Rehabilitation protocol without FES
- CIM-CON (Active Comparator): Each subject will receive 15 individual rehabilitation sessions, each lasting 60 minutes, conducted 3 to 5 times per week over a period of 5 to 3 weeks, depending on the weekly frequency,
  Intentional, repetitive movements, such as lower limb movements within goal-oriented mobility tasks (e.g., overground straight walking), will be performed without FES. The electrical stimulator will be positioned, and the amplitude will be set to zero
  Interventions: Other: Rehabilitation protocol without FES

INTERVENTIONS:
Other: Rehabilitation protocol: FES — Subjects diagnosed with CIP will follow the FES-based rehabilitation protocol
  Arms: CIP-FES
Other: Rehabilitation protocol without FES — Subjects belonging to the control group will follow the rehabilitation protocol without FES
  Arms: CIM-CON; CIP-CON
Other: Rehabilitation protocol: FES — Subjects diagnosed with CIM will follow the FES-based rehabilitation protocol
  Arms: CIM-FES

SUMMARY:
The aim of Re-Walk-Easy is to evaluate the effects of rehabilitation based on electrical stimulation on the motor performance of critically ill patients. The study will also investigate the pathophysiology of the two forms-the myopathic-predominant and the polyneuropathic-predominant variants-by examining the longitudinal progression of CIP and CIM and determining which form benefits more from electrical stimulation as a rehabilitative approach.

DETAILED DESCRIPTION:
Although rehabilitation is often recommended to patients with Intensive Care Unit Acquired Weakness (ICU-AW) to counteract the induced muscle weakness, systematic reviews failed to determine its efficacy. Neuro Muscular Electrical Stimulation (NMES) is part of clinical practice in ICU-AW however its effects are still under debate. The investigators hypothesize that this uncertainty stems from the lack of distinction between the two forms of the condition-Critical Illness Polyneuropathy (CIP) and Critical Illness Myopathy (CIM)-which have distinct pathological features and disease trajectories. In addition, the investigators hypothesize that motivating patients by requiring voluntary muscle activation during the Electrical Stimulation (i.e. Functional Electrical Stimulation - FES) will enhance rehabilitation.

The study will test the following hypothesis through a longitudinal clinical trial aimed at determining:

1. which form will benefit the most from FES based-rehabilitation,
2. the biomarkers of walking recovery in ICU-AW.

ELIGIBILITY:
Critical Illness Patient Inclusion Criteria:

* clinical diagnosis of tetra/paraparesis of peripheral origin as disclosed by ENG/EMG examination;
* be independent before the episode of critical illness

Critical Illness Patient Exclusion Criteria:

* history of previous comorbidity for ICU-AW;
* previous known chronic polyneuropathy;
* severe coagulopathy;
* severe disorder of consciousness;
* contraindications to Electrical Stimulation application

Healthy Subjects Exclusion Criteria:

* Prosthetic implants
* musculoskeletal, neurological, cardiovascular and pulmonary disorders that may alter the gait

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Medical Research Council - Sum Score (MRC-SS) | Baseline (T0), after 15 rehabilitation sessions (each session is 60 minutes, T2), 3-month follow-up (T3)
  The scale measures six bilateral muscle groups (wrist flexion, elbow flexion, shoulder abduction, ankle dorsiflexion, knee extension and hip flexion) with a maximum score of 60 points (normality) and a minimum score of 0 points (No muscle contraction visible or palpable).

SECONDARY OUTCOMES:
Walking velocity on 10 meters walking test | Baseline (T0), 3-week from T0 (T1), after 15 rehabilitation sessions (each session is 60 minutes, T2), 3-month follow-up (T3)
  Walking speed is measured by the timed 10-meter Walk Test (10MWT). Participants walk a distance of 10 meters at their usual speed with their usual walking aids. Participants are timed while walking 10 meters from a starting point to an end point. Time taken from meter 2 to meter 8. Two repetitions are completed and the average time is used to calculate walking speed in metres/second. During the test, EMG and kinematic data will be recorded using EMG-sensors and three IMUs, two placed on the feet and one on the lower back.
Modified Barthel Index | Baseline (T0), after 15 rehabilitation sessions (each session is 60 minutes, T2), 3-month follow-up (T3)
  Measurement instrument, based on an ordinal scale, commonly used to assess daily life activities. The total score ranges from 0 (total dependency) to 100 (full autonomy).
Instrumented Six Minute Walk Test | Baseline (T0), 3-week from T0 (T1), after 15 rehabilitation sessions (each session is 60 minutes, T2), 3-month follow-up (T3)
  Walking capacity is measured with the Participant timed while walking a 30 meter track constantly for 6 minutes. Participants are permitted to use their walking aids if necessary, and Patients will wear an IMU. The distance walked in 6 minutes is recorded and reported in meters.
Timed Up and Go Test | Baseline (T0), 3-week from T0 (T1), after 15 rehabilitation sessions (each session is 60 minutes, T2), 3-month follow-up (T3)
  The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk. Patient are timed while standing up from a chair walking 3 meters, turning around, walking 3 meters and sitting down again.
  The patient sits in the chair with his/her back against the chair back. On the command "go," the patient rises from the chair, walks 3 meters at a comfortable and safe pace, turns, walks back to the chair and sits down.
  Timing begins at the instruction "go" and stops when the patient is seated.
Euro Quality of Life-5 -dimension Questionnaire | Baseline (T0), after 15 rehabilitation sessions (each session is 60 minutes, T2), 3-month follow-up (T3)
  EQ-5D-5L is a standardized instrument for use as a measure of health for clinical and economic appraisal.Applicable to a wide range of health conditions and treatments, the EQ-5D health questionnaire provides a simple descriptive profile and a single index value for health status.
  Measures the 5 dimensions of:
  mobility self-care usual activities pain/discomfort anxiety/depression Each dimension is scored on a Likert scale of 5 levels, with higher scores indicating more severe problems.
Client Satisfaction Questionnaire - CSQ | After 15 rehabilitation sessions (each session is 60 minutes, T2)
  It measures the degree of satisfaction of the subject in terms of improvement of the treatment received. The total score ranges from 0 (not satisfied) to 40(full satisfied).
Needle Electromyography-based parameters | Baseline (T0), after 15 rehabilitation sessions (each session is 60 minutes, T2), 3-month follow-up (T3)
  Needle Electromyography (EMG) will be used for both qualitative and quantitative analysis of muscle activity.
  Collected data:
  1. Spontaneous activity: Analysis of fibrillation potentials and positive sharp waves in target muscles of the upper and lower limbs.
  2. Voluntary activity: Analysis of motor unit potential recruitment patterns and amplitude in target muscles of the upper and lower limbs.
Electroneurography (ENG) and Nerve Conduction Studies | Baseline (T0), after 15 rehabilitation sessions (each session is 60 minutes, T2), 3-month follow-up (T3)
  Electroneurography (ENG) data will be collected separately for motor and sensory nerve conduction studies. Direct muscle stimulation will be performed to differentiate predominantly neuropathic from predominantly myopathic forms. Collected data will be:
  1. Amplitude of Compound Muscle Action Potential (CMAP) (measured in millivolts [mV]).
  2. Amplitude of Sensory Nerve Action Potential (SNAP) (measured in millivolts [mV]).
Electroneurography (ENG) and Nerve Conduction Studies | Baseline (T0), after 15 rehabilitation sessions (each session is 60 minutes, T2), 3-month follow-up (T3)
  Electroneurography (ENG) data will be collected separately for motor and sensory nerve conduction studies. Direct muscle stimulation will be performed to differentiate predominantly neuropathic from predominantly myopathic forms. Collected data will be:
  1. Latency of CMAP (measured in milliseconds [ms]).
  2. Latency of SNAP (measured in milliseconds [ms]).
  3. Duration of CMAP(measured in milliseconds [ms]).
  4. Duration of SNAP (measured in milliseconds [ms]).
  5. F-response latency of major nerve trunks (measured in milliseconds [ms]).
Postural capabilities will be evaluated based on body kinetics | Baseline (T0), 3-week from T0 (T1), after 15 rehabilitation sessions (each session is 60 minutes, T2), 3-month follow-up (T3)
  Postural data of the lower limb will be acquired using an optoelectronic system combined with two force plates, sampling at 2000 Hz. Utilizing data processing techniques, deviations from normal postural dynamics will be determined.
Fall diary | From baseline (T0) to 3-month follow-up (T3)
  Falls diaries gather information about the frequency of falls and the circumstances in which the fall occurred. The information include: date/time of fall; location of fall; what caused the fall; type of injury sustained; action taken.
Report of adverse events | From baseline (T0) to post-treatment evaluation, after the 15 rehabilitation sessions (each session is 60 minutes, T2)
  Organized reporting of adverse events occurring during the use of the device

OTHER OUTCOMES:
Gender data | Baseline (T0)
  Gender of enrolled subject
Age data | Baseline (T0)
  Age of enrolled subject
Scholarity data | Baseline (T0)
  Scholarity of enrolled subject

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi Onlus, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Preliminary data will be available at the end of the study
Access Criteria: at request to the Principal investigator

REFERENCES:
- [Background] Van Lancker K, Bretz F, Dukes O. Covariate adjustment in randomized controlled trials: General concepts and practical considerations. Clin Trials. 2024 Aug;21(4):399-411. doi: 10.1177/17407745241251568. Epub 2024 Jun 2. PMID 38825841
- [Background] Dobkin BH. Progressive Staging of Pilot Studies to Improve Phase III Trials for Motor Interventions. Neurorehabil Neural Repair. 2009 Mar-Apr;23(3):197-206. doi: 10.1177/1545968309331863. PMID 19240197
- [Background] Gordon T. Electrical Stimulation to Enhance Axon Regeneration After Peripheral Nerve Injuries in Animal Models and Humans. Neurotherapeutics. 2016 Apr;13(2):295-310. doi: 10.1007/s13311-015-0415-1. PMID 26754579
- [Background] Jonsdottir J, Thorsen R, Aprile I, Galeri S, Spannocchi G, Beghi E, Bianchi E, Montesano A, Ferrarin M. Arm rehabilitation in post stroke subjects: A randomized controlled trial on the efficacy of myoelectrically driven FES applied in a task-oriented approach. PLoS One. 2017 Dec 4;12(12):e0188642. doi: 10.1371/journal.pone.0188642. eCollection 2017. PMID 29200424
- [Background] Perini G, Bertoni R, Thorsen R, Carpinella I, Lencioni T, Ferrarin M, Jonsdottir J. Sequentially applied myoelectrically controlled FES in a task-oriented approach and robotic therapy for the recovery of upper limb in post-stroke patients: A randomized controlled pilot study. Technol Health Care. 2021;29(3):419-429. doi: 10.3233/THC-202371. PMID 33386831
- [Background] Connolly B, O'Neill B, Salisbury L, McDowell K, Blackwood B; Enhanced Recovery After Critical Illness Programme Group. Physical rehabilitation interventions for adult patients with critical illness across the continuum of recovery: an overview of systematic reviews protocol. Syst Rev. 2015 Sep 29;4:130. doi: 10.1186/s13643-015-0119-y. PMID 26419458
- [Background] Mehrholz J, Pohl M, Kugler J, Burridge J, Muckel S, Elsner B. Physical rehabilitation for critical illness myopathy and neuropathy: an abridged version of Cochrane Systematic Review. Eur J Phys Rehabil Med. 2015 Oct;51(5):655-61. Epub 2015 Jul 9. PMID 26158919
- [Background] Liu M, Luo J, Zhou J, Zhu X. Intervention effect of neuromuscular electrical stimulation on ICU acquired weakness: A meta-analysis. Int J Nurs Sci. 2020 Mar 10;7(2):228-237. doi: 10.1016/j.ijnss.2020.03.002. eCollection 2020 Apr 10. PMID 32685621
- [Background] Garcia-Perez-de-Sevilla G, Sanchez-Pinto Pinto B. Effectiveness of physical exercise and neuromuscular electrical stimulation interventions for preventing and treating intensive care unit-acquired weakness: A systematic review of randomized controlled trials. Intensive Crit Care Nurs. 2023 Feb;74:103333. doi: 10.1016/j.iccn.2022.103333. Epub 2022 Oct 22. PMID 36283894
- [Background] Wang W, Xu C, Ma X, Zhang X, Xie P. Intensive Care Unit-Acquired Weakness: A Review of Recent Progress With a Look Toward the Future. Front Med (Lausanne). 2020 Nov 23;7:559789. doi: 10.3389/fmed.2020.559789. eCollection 2020. PMID 33330523
- [Background] Latronico N, Bolton CF. Critical illness polyneuropathy and myopathy: a major cause of muscle weakness and paralysis. Lancet Neurol. 2011 Oct;10(10):931-41. doi: 10.1016/S1474-4422(11)70178-8. PMID 21939902